CLINICAL TRIAL: NCT01679834
Title: A Roche Project in Cooperation With the Bng (Association of German Resident Gastroenterologists) for Quality Assurance in the Dual- or Triple-therapy of Chronic Hepatitis C With Peg-(40kd)-Interferon Alfa 2a (Pegasys) at Hepatology Centers
Brief Title: An Observational Study of Pegasys in Dual- or Triple-Therapy in Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25724
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, observational study will assess the efficacy and the safety of Pegasys (peginterferon alfa 2a) in dual- or triple therapy in patients with chronic hepatitis C. Patients will receive Pegasys and/or ribavirin and/or a protease inhibitor according to local guidelines. Data will be collected for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of chronic hepatitis C
* Patients receiving treatment with Pegasys and/or Copegus (ribavirin) and/or a protease inhibitor according to local label

Exclusion Criteria:

* Contraindications against Pegasys or Copegus
* Not willing or unable to sign written informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C infection
Sampling Method: Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2014-11-24 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 24 weeks after end of treatment

SECONDARY OUTCOMES:
Rapid virological response | 4 weeks after start of treatment
Early Virological Response | 12 weeks after start of treatment
Safety: incidence of adverse events | up to 24 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Germany (2):
  - Hanover
  - Herne